CLINICAL TRIAL: NCT04386291
Title: Meditation and Yoga for Heightened Anxiety Related to COVID-19
Brief Title: Meditation and Kundalini Yoga for Heightened Anxiety Related to COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Brian A Fallon, Professor of Psychiatry, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7987
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Generalized Anxiety; Health Anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three treatment arms: Anxiety Reduction Training (A.R.T.), ART with Kundalini Yoga, ART with Meditation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anxiety Reduction Training (A.R.T.) (Active Comparator): Participants will received biweekly on-line lessons that provide education and strategies to reduce stress and disturbing thoughts and improve healthy coping and sleep. .
  Interventions: Behavioral: Anxiety Reduction Training
- ART and Kundalini Yoga (Experimental): This combines ART with a daily 30 minute practice of Kundalini Yoga (stretching, guided breathing, and meditation). Accessible by smart phone, tablet or computer.
  Interventions: Behavioral: Anxiety Reduction Training; Behavioral: Kundalini Yoga and Anxiety Reduction Training
- ART and Meditation (Experimental): This combines ART with a daily 15 minute meditation with stress reduction techniques and guided breathing.
  Interventions: Behavioral: Anxiety Reduction Training; Behavioral: Meditation and Anxiety Reduction Training

INTERVENTIONS:
Behavioral: Anxiety Reduction Training — Educational material will be provided every two weeks that address different aspects of anxiety and cognitive-behavioral approaches to reduce anxiety and stress.
Behavioral: Kundalini Yoga and Anxiety Reduction Training — Daily practice of Kundalini Yoga (light stretching, breathing exercises, and meditation) guided by on-line video instruction, as well as the biweekly anxiety reduction psychoeducation.
  Arms: ART and Kundalini Yoga
Behavioral: Meditation and Anxiety Reduction Training — Daily practice of meditation (muscle relaxation, breathing, and meditation) guided by on-line video instruction, as well as the biweekly anxiety reduction psychoeducation.
  Arms: ART and Meditation

SUMMARY:
This randomized clinical on-line study examines whether whether a daily practice of meditation or Kundalini Yoga with anxiety reduction training leads to a greater reduction in anxiety than anxiety reduction training alone.

DETAILED DESCRIPTION:
The individual and societal costs of the COVID-19 pandemic are wide-ranging. Based on past epidemics and on emerging data, anxiety and depression rates will increase, along with anger, grief, somatic complaints, and post-traumatic stress. Coping skills will be challenged, particularly as anxiety, uncertainty, and personal loss increase.

While anxiety is a healthy response to danger, excessive anxiety can be debilitating and impair our coping skills. Illness anxiety may also increase given concerns about infection risks to self and others.

This randomized on-line study is for individuals with anxiety and distress triggered by COVID-19 who have not yet been infected with the novel corona virus. .

The primary study goal is to examine the extent to which anxiety can be reduced through the use of on-line training programs. All participants will receive Anxiety Reduction Training using cognitive-behavioral methods known to be helpful in reducing stress, anxiety, depression, and insomnia. In addition, two-thirds of participants will be randomly assigned to receive training in either Kundalini Yoga (KY) or mindfulness meditation. The investigators will assess the degree to which each of these training programs lead to reduced stress, improved well-being, decreased multisystem symptoms, enhanced mood, and reduced cognitive complaints. Participants will complete self-report assessments at 2-week intervals during the 8 weeks of the acute phase of the study and then again 3- and 6-months later.

The current study may reveal that addressing emergent anxiety early through online self-guided treatment approaches can lead to improved short- and long-term outcome. Findings from this study may reveal that these inexpensive easily disseminated on-line programs can be helpful to enhance coping and improve mental health in the context of large-scale public health crises.

ELIGIBILITY:
Inclusion Criteria:

1. Heightened anxiety triggered or exacerbated by COVID-19
2. Anxiety it least mild-moderate in severity
3. English speaking and living in the United States
4. Access to a smart phone, tablet, or computer with internet
5. Able to read and understand English

Exclusion Criteria:

1. Individuals with severe depression or substance abuse
2. Individuals with a current or past history of psychosis, bipolar disorder, or PTSD.
3. Individuals with physical disability that might make study participation difficult.
4. Individuals with an unstable medical illness or a history of cardiac disease
5. Individuals with a current daily practice of meditation or Kundalini yoga
6. Individuals with confirmed or suspected COVID-19
7. Individuals who are currently pregnant or anticipate being pregnant during study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2022-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Fallon, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - ProofPilot (Virtual Study: https://proofpilot.com/covid-anxiety/), New York, New York
  - Columbia University Department of Psychiatry, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlson LE, Garland SN. Impact of mindfulness-based stress reduction (MBSR) on sleep, mood, stress and fatigue symptoms in cancer outpatients. Int J Behav Med. 2005;12(4):278-85. doi: 10.1207/s15327558ijbm1204_9. PMID 16262547
- [Background] Grossman P, Kappos L, Gensicke H, D'Souza M, Mohr DC, Penner IK, Steiner C. MS quality of life, depression, and fatigue improve after mindfulness training: a randomized trial. Neurology. 2010 Sep 28;75(13):1141-9. doi: 10.1212/WNL.0b013e3181f4d80d. PMID 20876468
- [Background] Khalsa MK, Greiner-Ferris JM, Hofmann SG, Khalsa SB. Yoga-enhanced cognitive behavioural therapy (Y-CBT) for anxiety management: a pilot study. Clin Psychol Psychother. 2015 Jul-Aug;22(4):364-71. doi: 10.1002/cpp.1902. Epub 2014 May 7. PMID 24804619
- [Background] Shannahoff-Khalsa D, Fernandes RY, Pereira CAB, March JS, Leckman JF, Golshan S, Vieira MSR, Polanczyk GV, Miguel EC, Shavitt RG. Kundalini Yoga Meditation Versus the Relaxation Response Meditation for Treating Adults With Obsessive-Compulsive Disorder: A Randomized Clinical Trial. Front Psychiatry. 2019 Nov 11;10:793. doi: 10.3389/fpsyt.2019.00793. eCollection 2019. PMID 31780963
- [Background] Wang YY, Li XH, Zheng W, Xu ZY, Ng CH, Ungvari GS, Yuan Z, Xiang YT. Mindfulness-based interventions for major depressive disorder: A comprehensive meta-analysis of randomized controlled trials. J Affect Disord. 2018 Mar 15;229:429-436. doi: 10.1016/j.jad.2017.12.093. Epub 2018 Jan 3. PMID 29331704
- [Background] Kladnitski N, Smith J, Uppal S, James MA, Allen AR, Andrews G, Newby JM. Transdiagnostic internet-delivered CBT and mindfulness-based treatment for depression and anxiety: A randomised controlled trial. Internet Interv. 2020 Feb 13;20:100310. doi: 10.1016/j.invent.2020.100310. eCollection 2020 Apr. PMID 32140427
- [Background] Andersson E, Enander J, Andren P, Hedman E, Ljotsson B, Hursti T, Bergstrom J, Kaldo V, Lindefors N, Andersson G, Ruck C. Internet-based cognitive behaviour therapy for obsessive-compulsive disorder: a randomized controlled trial. Psychol Med. 2012 Oct;42(10):2193-203. doi: 10.1017/S0033291712000244. Epub 2012 Feb 21. PMID 22348650
- [Background] Spijkerman MP, Pots WT, Bohlmeijer ET. Effectiveness of online mindfulness-based interventions in improving mental health: A review and meta-analysis of randomised controlled trials. Clin Psychol Rev. 2016 Apr;45:102-14. doi: 10.1016/j.cpr.2016.03.009. Epub 2016 Apr 1. PMID 27111302

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
Started | 83 | 88 | 85
Completed | 21 | 12 | 23
Not Completed | 62 | 76 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation | Total
Number analyzed (Participants) | 83 | 88 | 85 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.4) | 45.6 (12.7) | 49.6 (13.3) | 47.4 (13.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 72 | 81 | 75 | 228
  Male | 11 | 6 | 10 | 27
  Transgender | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 3 | 7
  White | 77 | 74 | 74 | 225
  More than one race | 1 | 5 | 4 | 10
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 83 | 88 | 85 | 256

OUTCOME MEASURES:

1. Primary Outcome: GAD-7
Description: Generalized Anxiety Disorder 7-item scale (range 0-21, higher score indicates more pronounced anxiety). A change score is calculated based on baseline score minus week 8 score.
Time Frame: 8 weeks
Population: Analysis of a change score between baseline and week 8 for those who those who were randomized into one of the study arms and completed active treatment phase. A larger positive change score indicates a greater improvement on a scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
Number analyzed (Participants) | 14 | 6 | 16
score on a scale | 4.7 (4.4) | 7.8 (2.9) | 4.9 (4.6)
Statistical Analysis 1: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Kundalini Yoga; Test type: Superiority; p = 0.071, t-test, 1 sided; Mean Difference (Final Values) = -1.54
Statistical Analysis 2: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Meditation; Test type: Superiority; p = 0.46, t-test, 1 sided; Mean Difference (Final Values) = -0.09

2. Primary Outcome: Whiteley 8
Description: Health Anxiety 8-item scale (range 0-32, higher score indicates more pronounced anxiety). A change score is calculated based on baseline score minus week 8 score.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
Number analyzed (Participants) | 21 | 12 | 23
score on a scale | 0.05 (4.9) | 3.9 (3.4) | 2.5 (4.5)
Statistical Analysis 1: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Kundalini Yoga; Test type: Superiority; p = 0.01, t-test, 1 sided; Mean Difference (Final Values) = -2.4
Statistical Analysis 2: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Meditation; Test type: Superiority; p = 0.04, t-test, 1 sided; Mean Difference (Final Values) = -1.76

3. Secondary Outcome: PHQ-8
Description: Patient Health Questionnaire 8 - an 8 item measure of depression (range 0-24, higher score indicates more pronounced depression). A change score is calculated based on baseline score minus week 8 score.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
Number analyzed (Participants) | 13 | 6 | 15
score on a scale | 4.8 (3.7) | 7.8 (5.3) | 4.5 (6.1)
Statistical Analysis 1: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Kundalini Yoga; Test type: Superiority; p = 0.08, t-test, 1 sided; Mean Difference (Final Values) = -1.47
Statistical Analysis 2: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Meditation; Test type: Superiority; p = 0.5, t-test, 1 sided; Mean Difference (Final Values) = 0.12

4. Secondary Outcome: SS-8
Description: Somatic Symptom Scale-8 an 8-item measure of symptom burden (range 0-32, higher score represents worsening of somatic symptoms). A change score is calculated based on baseline score minus week 8 score.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
Number analyzed (Participants) | 21 | 12 | 23
score on a scale | -3.8 (4.4) | -2.8 (4.1) | -1.7 (4.5)
Statistical Analysis 1: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Kundalini Yoga; Test type: Superiority; p = 0.25, t-test, 1 sided; Mean Difference (Final Values) = -0.68
Statistical Analysis 2: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Meditation; Test type: Superiority; p = 0.065, t-test, 1 sided; Mean Difference (Final Values) = -1.54

5. Secondary Outcome: Applied Cognition 1.0
Description: An 8-item self-report measure of cognitive function (range 8-40, higher is better). A change score is calculated based on baseline score minus week 8 score.
Time Frame: 8 weeks
Population: Analysis of a change score between baseline and week 8 for those who those who were randomized into one of the study arms and completed active treatment phase. A larger negative change score indicates a greater improvement on a scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
Number analyzed (Participants) | 21 | 11 | 21
score on a scale | -4.1 (5.5) | -6.6 (5.5) | -5.1 (6.5)
Statistical Analysis 1: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Kundalini Yoga; Test type: Superiority; p = 0.88, t-test, 1 sided; Mean Difference (Final Values) = 1.24
Statistical Analysis 2: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Meditation; Test type: Superiority; p = 0.7, t-test, 1 sided; Mean Difference (Final Values) = 0.56

6. Secondary Outcome: PROMIS-4 Sleep Disturbance
Description: A 4-item self-report assessment of sleep disturbance (range 4-20, higher score indicates more sleep disturbance). A change score is calculated based on baseline score minus week 8 score.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
Number analyzed (Participants) | 21 | 11 | 23
score on a scale | 1.5 (3.0) | 3.7 (3.8) | 3.3 (4.3)
Statistical Analysis 1: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Kundalini Yoga; Test type: Superiority; p = 0.038, t-test, 1 sided; Mean Difference (Final Values) = -1.84
Statistical Analysis 2: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Meditation; Test type: Superiority; p = 0.059, t-test, 1 sided; Mean Difference (Final Values) = -1.59

7. Secondary Outcome: ERQ
Description: Emotional Regulation Questionnaire - a 10-item measure of emotional regulation; the reappraisal subscale has a range: of 6-42, higher score reflects improvement; while the suppression subscale has a range of 4-28, higher score considered worsening status. A change score is calculated based on baseline score minus week 8 score.
Time Frame: 8 weeks
Population: Analysis of a change score between baseline and week 8 for those who those who were randomized into one of the study arms and completed active treatment phase. A larger negative change score on the reappraisal subscale indicates a greater improvement on a scale. A larger positive change score on the suppression subscale indicates a greater improvement on a scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
Number analyzed (Participants) | 21 | 11 | 23
score on a scale
  Reappraisal Subscale | -1.9 (4.7) | -5.5 (7.8) | -2.9 (6.3)
  Suppression Subscale | -16.2 (8.1) | -13.9 (9.1) | -16.5 (8.9)
Statistical Analysis 1: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Kundalini Yoga; Reappraisal subscale analysis; Test type: Superiority; p = 0.9, t-test, 1 sided; Median Difference (Final Values) = 1.58
Statistical Analysis 2: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Kundalini Yoga; Subpression subscale analysis; Test type: Superiority; p = 0.23, t-test, 1 sided; Mean Difference (Net) = -0.73
Statistical Analysis 3: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Meditation; Reappraisal subscale analysis; Test type: Superiority; p = 0.7, t-test, 1 sided; Mean Difference (Final Values) = 0.54
Statistical Analysis 4: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Meditation; Suppression subscale analysis; Test type: Superiority; p = 0.5, t-test, 1 sided; Mean Difference (Final Values) = 0.1

8. Secondary Outcome: Perceived Stress Scale
Description: A 10-item scale assessing the perception of events in one's life as stressful (0-40, higher score indicates more pronounced perception of stress).A change score is calculated based on baseline score minus week 8 score.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
Number analyzed (Participants) | 21 | 11 | 22
score on a scale | 4.1 (6.5) | 6.0 (5.9) | 6.5 (8.1)
Statistical Analysis 1: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Kundalini Yoga vs ART and Meditation; Test type: Superiority; p = 0.5, ANOVA; Mean Difference (Final Values) = 0.67

9. Secondary Outcome: Brief Hypervigilance Scale
Description: A 5-item scale assessing hypervigilance (0-20, higher score indicates greater hypervigilance). A change score is calculated based on baseline score minus week 8 score.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
Number analyzed (Participants) | 21 | 11 | 22
score on a scale | 1.2 (2.4) | 3.5 (4.1) | 0.4 (3.2)
Statistical Analysis 1: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Kundalini Yoga; Test type: Superiority; p = 0.076, Wilcoxon (Mann-Whitney); Mann-Witney was used because assumption of normality of variance was violated; mean rank difference = 79.0
Statistical Analysis 2: Comparison: Anxiety Reduction Training (A.R.T.) vs ART and Meditation; Test type: Superiority; p = 0.8, t-test, 1 sided; Mean Difference (Final Values) = 0.9

ADVERSE EVENTS:
Time Frame: 8 weeks of acute treatment phase
Description: Adverse events information was collected via online platform at baseline and 8 weeks with a Healthcare Utilization questionnaire. Questions addressed adverse experiences and overnight hospitalizations. In addition, participants could reach out to research team if they experienced any distress with their program of treatment.
Arm/Group | Anxiety Reduction Training (A.R.T.) | ART and Kundalini Yoga | ART and Meditation
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/88 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/88 | 0/85
Other Adverse Events (participants affected / at risk) | 0/83 | 0/88 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT04386291/Prot_SAP_000.pdf